CLINICAL TRIAL: NCT02110862
Title: Scintigraphic Evaluation of IPAA Function in CU Patients
Brief Title: Scintigraphic Evaluation of IPAA Function in Patients With Ulcerative Colitis
Acronym: SKIPO
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mie Dilling Kjaer, MD, Odense University Hospital
Other Study IDs: Skipo-2013; S-20110117 (Other: The National Committee on Health Research Ethics Denmark)
Record Dates: First submitted 2013-04-30; First posted 2014-04-10 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ulcerative colitis patients with ileal-pouch-anal anastomosis
  Interventions: Other: Transittime. Defecography

INTERVENTIONS:
Other: Transittime. Defecography

SUMMARY:
The aim of this study is to evaluate scintigraphic methods as objective factors for functional outcome in patients treated with ileal-pouch-anal anastomosis (IPAA). The gastrointestinal transit-time and the degree of evacuation are evaluated in relation to the functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulcerative colitis
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit-time | 12 weeks
  The small bowel transittime until food is in the IPAA

CONTACTS AND LOCATIONS:
Overall Officials: Mie Kjaer, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark